CLINICAL TRIAL: NCT03329534
Title: Mechanisms Underlying Development of Barrett's Esophagus in Patients With Gluten Related Disorders
Brief Title: Gluten Related Disorders in Barrett's Esophagus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GRD in BE
Record Dates: First submitted 2017-10-18; First posted 2017-11-06 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2017-10

CONDITIONS: Celiac Disease; Barrett Esophagus; Gluten Sensitivity; GERD
MeSH Terms: conditions — Celiac Disease; Barrett Esophagus; Gastroesophageal Reflux | interventions — Diet, Gluten-Free

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects with GRDs (Experimental): An intervention of a change in diet, specifically a gluten free diet taught by a health care professional will be administered for one month's time.
  Interventions: Other: Gluten free diet
- Subjects without GRDs (Active Comparator): An intervention of a change in diet, specifically a gluten free diet taught by a health-care professional will be administered for one month's time.
  Interventions: Other: Gluten free diet

INTERVENTIONS:
Other: Gluten free diet — A month long gluten free diet

SUMMARY:
In a small group of people gluten, a storage protein commonly in wheat and other grains, can cause gut inflammation and symptoms like diarrhea and abdominal pain. Gluten-related disorders include celiac disease (CD) and non-celiac gluten sensitivity (NCGS) and are treated by starting a gluten free diet (GFD). Patients with CD and NCGS also more commonly experience esophageal reflux and damage to the lining of the esophagus. A potential consequence of long-standing heartburn is Barrett's esophagus (BE), a major risk factor for cancer of the esophagus.

This study aims to investigate the mechanism that leads to reflux and BE in those with gluten related disorders, and to assess if a GFD is beneficial. We will study the upper gut function and reflux activity in patients with BE both with and without a GRD disorder. Testing will occur before and after a gluten free diet is instituted. The results will help inform health care providers and patients about the connection between gluten-related disorders, reflux, BE, and the role of GFD.

DETAILED DESCRIPTION:
Perhaps patient's with gluten related disorders develop Barrett's esophagus due to non-acid reflux precipitated by upper gastrointestinal motility changes that respond to a gluten free diet; whereas patients without gluten related disorders develop Barrett's due to the accepted mechanism of acid reflux.

The primary objectives are to explore if patients with gluten-related disorders (CD and GS) may have an altered mechanism of developing Barrett's esophagus typified by increased alkali reflux compared to those without gluten-related disorders; and to determine if this mechanism (altered motility and increased non-acid reflux) responds to a gluten free diet.

Specific objectives include assessing whether patients with GRD and Barrett's esophagus have altered esophageal reflux extent, frequency, and type (assessed by pH-impedance); altered symptom profiles; differential esophageal body and sphincter pressures (assessed by manometry); aberrant gastroduodenal motility (assessed by videofluoroscopy) in comparison to patients with BE and no GRD. Finally a gluten free diet will be instituted to assess whether a gluten-free diet alters esophageal reflux extent, frequency, and type or symptom profiles in those with BE with and without a GRD.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and over
* Barrett's Esophagus diagnosis based on endoscopy and esophageal biopsies
* Patients able to comply to the study procedures, according to the investigator's own judgment

Exclusion Criteria:

* Patients who have been on a gluten free diet within the last six months
* History of bariatric surgery, fundoplication, or gastrectomy (partial or complete)
* Connective tissue disease
* Concurrent organic GI pathology other than benign polyps, haemorrhoids, lipomas, H. pylori infection, diverticulosis, and melanosis coli
* Chronic treatment with high dose opioids
* Alcohol or drug abuse
* Pregnant or breastfeeding women. Women enrolling in the study will be advised to avoid pregnancy during the course of the study by using adequate birth control such as abstinence, oral contraceptive pill, barrier contraceptives (i.e condom). If a subject becomes pregnant she will be withdrawn from the study.
* Concurrent systemic disease and/or laboratory abnormalities considered by investigators to be a risk or that could interfere with data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Ratio of non-acidic to acidic reflux events | At study start and at one month after a gluten free diet
  Proportion of non-acid to acid reflux events as determined by pH-impedance

SECONDARY OUTCOMES:
Reflux disease questionnaire | At study start and one month after a gluten free diet
  12 questions with six choices each. Results are added such that best score is 12 and worst score is 72.
Esophageal motility | At study start
  Manometric findings of the upper and lower sphincters and esophageal body
Upper gastrointestinal motility | At study start
  Fluoroscopic findings of gastroduodenal motility
Leeds short form questionnaire | At study start and one month after a gluten free diet
  Questionnaire for dyspepsia. Nine questions with five choices each. Only eight question scores are summed. Best score is 8 and worst score is 40.
Gastroesophageal reflux disease-health related quality of life instrument | At study start and one month after a gluten free diet
  11 questions. Ten of them are summed with six choices each. The best score is 0 and the worst score is 50.

CONTACTS AND LOCATIONS:
Overall Officials: Premysl Bercik, MD, Study Director — McMaster University

IPD SHARING:
Plan to Share IPD: No